CLINICAL TRIAL: NCT03598933
Title: Cricopharyngeal Dysfunction in Adults: Diagnostic and Therapeutic Effects of Cricopharyngeal Botulinum Toxin (Botox) Injection
Brief Title: Cricopharyngeal Dysfunction in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7053
Record Dates: First submitted 2018-07-11; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Upper Esophageal Sphincter
Keywords: Upper Esophageal Sphincter; botulinum toxin; Cricopharyngeal dysfunction; Cricopharyngeal botulinum toxin injection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study, after reviewing the recent literature, is to corroborate the thesis of the authors considering the injection of botulinum toxin as a gesture that is both diagnostic and therapeutic in the disorders of the Upper Esophageal Sphincter and reinforce the results already published with a larger series of patients.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman whose age older than 18 years
* Dysphagia with solids and / or liquids
* Dysfunction of primary or secondary Upper Esophageal Sphincter with indirect video-fibroscopy and / or video-fluoroscopy and / or high resolution pharyngo-oesophageal manometry
* Subject having at least one injection of botulinum toxin A in the crico-pharyngeal muscle for Upper Esophageal Sphincter dysfunction in the ENT department and cervico-facial surgery of Hautepierre.
* Subject who has consented to the use of his data from his medical file for the purpose of this research

Exclusion Criteria:

* Myotomy in the first place
* Refusal of the subject to participate in the study
* Subject under the protection of justice
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Subject having at least one injection of botulinum toxin A in the crico-pharyngeal muscle for Upper Esophageal Sphincter dysfunction in the ENT department and cervico-facial surgery of Hautepierre.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Deglutition Handicap Index | The period from January 1st, 2017 to December 31st, 2017 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Schultz, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service ORL et chirurgie cervico-faciale, Strasbourg, France